CLINICAL TRIAL: NCT00497354
Title: Does a Low Volume Ultrasound-Guided Technique Reduce Common Complications of Interscalene Brachial Plexus Block?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SHSCA01
Record Dates: First submitted 2007-07-03; First posted 2007-07-06 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Pain After Shoulder Surgery
Keywords: Ultrasound, Complications, Regional Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Variation in volume of local anesthetic
Procedure: Ultrasound-guided interscalene brachial plexus block

SUMMARY:
Peripheral nerve blocks provide many advantages for patients (excellent pain control and reduction in nausea) undergoing upper and lower limb surgery however several commonly occurring complications can produce annoying but sometimes serious adverse effects. The interscalene brachial plexus block (ISBPB) is one such technique, commonly performed for shoulder surgery, but also produces paralysis of the diaphragm, Horner's syndrome and sometimes vocal cord paralysis with standard volumes of local anesthetic. This threat of these side effects limits the use of ISBPB in many patients who would particularly benefit e.g. patients with lung disease. Recently the use of ultrasound guidance is allowing practitioners to place smaller volumes of local anesthetic with much greater accuracy. This can potentially avoid anesthetizing important adjacent nerves to the target structure. If ultrasound-guided techniques with smaller volumes of local anesthetic could be demonstrated to reduce the incidence of complications without reducing effectiveness this would be very beneficial for patients.This will be the first randomized, double blind study to evaluate if an ultrasound-guided ISBPB with low volumes of local anesthetic can reduce complications for patients whilst maintaining quality of anesthesia and pain relief in the intra-operative and postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective shoulder surgery.
* Patients aged >=18 and <=70 years
* ASA I-III
* BMI<35

Exclusion Criteria:

* Preexisting COPD
* Unstable asthma
* Psychiatric history
* Allergy to ropivacaine.
* Opioid tolerance (>30mg oral morphine or equivalent/day)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2007-07; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic paresis | 30 minutes post block insertion

SECONDARY OUTCOMES:
Analgesic efficacy | 30,60,90,120 minutes post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Colin JL McCartney, FRCA, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada